CLINICAL TRIAL: NCT06607224
Title: Effect of the Use of Continuous Glucose Monitoring Versus Standard Glycemic Control for Insulin Therapy Adjustment and Decision Making in Noncritical Patients with Type 2 Diabetes Hospitalized in Medical and Surgical Wards.
Brief Title: Effect of the Use of Continuous Glucose Monitoring Versus Standard Glycemic Control in Hospitalized Patients with Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Olga Gonzalez Albarran, Principal Investigator, PhD, MD, Specialist in Endocrinology, Hospital General Universitario Gregorio Marañon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ENDO2021-1
Record Dates: First submitted 2024-09-05; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus Type 2; Hospitalization
Keywords: continuous glucose monitoring; hyperglycemia; FreeStyle; Hospitalization; Time in range
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decision making guided by CGM (Experimental): Hospitalized patients with T2D in non-critical medical and surgical wards. The participants use FreeStyle 2-CGM and therapeutic decisions will be made based on CGM and GC parameters; with the presence of alarms for hypoglycemia or hyperglycemia activated for timely action. Blinded will be applied to patients; while the data will be open to the physicians in charge of the research in order to make daily modifications of insulin therapy. The CG controls will be of 6 points (before each meal and two hours after meals) with a standard Abbott FreeStyle Optium Neo glucometer. Basal-bolus scheme with basal insulin Glargine U-100 and prandial insulin Aspart will be used. Daily adjustments will be made based on protocol based of our department according to the international guidelines and previous research
  Interventions: Device: Experimental (Decision making guided by CGM)
- Decision making guided by CG (No Intervention): Hospitalized patients with T2D admitted in non-critical medical and surgical wards. The participants use FreeStyle 2-CGM with deactivated alarms. Blind will be applied for patients, nurses and physicians in charge of the investigation. Concomitant 6-point CG controls will be performed (before each meal and two hours after meals) with Abbott FreeStyle Optium Neo glucometer. Insulin therapy adjustments will be carried out by GC only. The CGM values in this group will be evaluated a posteriori. Basal-bolus schedule with basal insulin Glargine U-100 and prandial insulin Aspart will be used. Daily adjustments will be made based on protocols of our department according to the international guidelines.

INTERVENTIONS:
Device: Experimental (Decision making guided by CGM) — Patients use FSL2 and a smartphone. Libreview app will be used to assess interstitial glucose, alarms, and trend arrows, and LibreLinkUp app for research team. Concurrently, CG will be performed using the FreeStyle Optium Neo glucometer from Abbott. The nursing staff will be trained to manage and respond to alarms and trend arrows according to established protocols. The basal insulin adjustment protocol establishes with fasting and premeal targets between 140-180 mg/dL. For prandial insulin, corrective guidelines set according to each patient sensitivity factor, with additional adjustments for the intervention group based on trend arrows. The hypoglycemia alarm sets below 85 mg/dL. If activated, nursing staff will confirm the value via CG. If values are below 70 mg/dL, follow hypoglycemia protocol and if below 100 mg/dL with a descending trend arrow, 15 grams of slow-acting carbs. The hyperglycemia alarm will be set above 300 mg/dL and nurse inform investigators to make decisions.
  Other Names: CGM
  Arms: Decision making guided by CGM

SUMMARY:
Type 2 diabetes (T2D) is a common pathology in hospitalized patients and is associated with multiple comorbidities. Moreover, it is widely known that glycemic excursions increase hospital stay, infections, morbidity and mortality. Likewise, asymptomatic hypoglycemia and stress hyperglycemia in hospitalized patients is more frequent due to intercurrent pathology, medication, alteration of counter-regulatory hormones. Therefore, the use of continuous glucose monitoring (CGM) systems would be very useful as it allows early recognition of glycemic excursions and thus improve the management of insulin therapy. The primary objective is to demonstrate the increase in time in range (TIR) with the use of CGM for insulin therapy adjustment in hospitalized patients with T2D during their admission. The investigators randomized, parallel group, 2-arm, 40 participants; 20 in each group, patients with diagnosis of T2D prior to admission.

DETAILED DESCRIPTION:
Over the past few decades advances in diabetes technology have revolutionized patient care and metabolic control. The use of CGM has demonstrated substantial benefits on glycemic control in ambulatory patients compared to standard capillary blood glucose (CG) monitoring. However, in hospitalized patients, limitations on its use persist due to the lack of standardization of the data provided by CGM.

The use of CG has been the mainstay for monitoring and adjusting the treatment of hospitalized patients with diabetes. In the management for inpatients this test is commonly performed 3 to 4 times a day. However, this provides significant limitations due to its intermittent nature and the associated time burden for hospital nursing and ancillary staff for its determination.

Several studies have demonstrated that CGM detects more hyperglycemia and hypoglycemia in critically ill and non-critically ill patients. These studies have provided important information on patterns of glycemic control, with emphasis on early detection of glycemic excursions. However, there is still a need for further research to determine the efficacy of their use in glycemic adjustment, reliability in the hospital setting, and standardized protocols for their implementation and decision-making.

HYPOTHESIS The use of CGM allows an increase in TIR and improves the detection of clinically significant hypoglycemia and hyperglycemia in patients with T2D hospitalized on basal-bolus insulin therapy versus standard CG.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Admitted to medical or surgical wards with an expected hospitalization duration of more than 72 hours
* Requiring basal-bolus insulin therapy during hospitalization.

Exclusion Criteria:

* Pregnant women
* Severe mental illnesses
* Chronic use of high doses of ascorbic acid (equivalent to more than 500mg/day)
* Patients hospitalized in Intensive Care Units
* Severe cognitive impairment
* Prior outpatient CGM use
* Refusal of informed consent
* Patients on prolonged absolute diets or receiving artificial nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
The primary objective is to demonstrate the increase in TIR with the use of CGM for insulin therapy adjustment in hospitalized patients with T2D during their admission. | The days of sensor use during hospitalization (from 3 to 14 days).
  -Time in range (TIR) reported at the end of sensor use: results will be expressed in percentages and levels greater than 70% will be considered good glycemic control.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year
Access Criteria: 1 year
URL: https://saludanv.salud.madrid.org/hospitales/hgugm/Paginas/default.aspx

REFERENCES:
- [Background] Spanakis EK, Urrutia A, Galindo RJ, Vellanki P, Migdal AL, Davis G, Fayfman M, Idrees T, Pasquel FJ, Coronado WZ, Albury B, Moreno E, Singh LG, Marcano I, Lizama S, Gothong C, Munir K, Chesney C, Maguire R, Scott WH, Perez-Guzman MC, Cardona S, Peng L, Umpierrez GE. Continuous Glucose Monitoring-Guided Insulin Administration in Hospitalized Patients With Diabetes: A Randomized Clinical Trial. Diabetes Care. 2022 Oct 1;45(10):2369-2375. doi: 10.2337/dc22-0716. PMID 35984478
- [Background] Fortmann AL, Spierling Bagsic SR, Talavera L, Garcia IM, Sandoval H, Hottinger A, Philis-Tsimikas A. Glucose as the Fifth Vital Sign: A Randomized Controlled Trial of Continuous Glucose Monitoring in a Non-ICU Hospital Setting. Diabetes Care. 2020 Nov;43(11):2873-2877. doi: 10.2337/dc20-1016. Epub 2020 Aug 27. PMID 32855160
- [Background] Burt MG, Roberts GW, Aguilar-Loza NR, Stranks SN. Brief report: Comparison of continuous glucose monitoring and finger-prick blood glucose levels in hospitalized patients administered basal-bolus insulin. Diabetes Technol Ther. 2013 Mar;15(3):241-5. doi: 10.1089/dia.2012.0282. Epub 2013 Jan 29. PMID 23360391
- [Background] Wallia A, Umpierrez GE, Rushakoff RJ, Klonoff DC, Rubin DJ, Hill Golden S, Cook CB, Thompson B; DTS Continuous Glucose Monitoring in the Hospital Panel. Consensus Statement on Inpatient Use of Continuous Glucose Monitoring. J Diabetes Sci Technol. 2017 Sep;11(5):1036-1044. doi: 10.1177/1932296817706151. Epub 2017 Apr 21. PMID 28429611
- [Background] Umpierrez GE, Klonoff DC. Diabetes Technology Update: Use of Insulin Pumps and Continuous Glucose Monitoring in the Hospital. Diabetes Care. 2018 Aug;41(8):1579-1589. doi: 10.2337/dci18-0002. Epub 2018 Jun 23. PMID 29936424
- [Background] Gomez AM, Umpierrez GE, Munoz OM, Herrera F, Rubio C, Aschner P, Buendia R. Continuous Glucose Monitoring Versus Capillary Point-of-Care Testing for Inpatient Glycemic Control in Type 2 Diabetes Patients Hospitalized in the General Ward and Treated With a Basal Bolus Insulin Regimen. J Diabetes Sci Technol. 2015 Aug 31;10(2):325-9. doi: 10.1177/1932296815602905. PMID 26330394
- [Background] Spanakis EK, Cook CB, Kulasa K, Aloi JA, Bally L, Davis G, Dungan KM, Galindo RJ, Mendez CE, Pasquel FJ, Shah VN, Umpierrez GE, Aaron RE, Tian T, Yeung AM, Huang J, Klonoff DC. A Consensus Statement for Continuous Glucose Monitoring Metrics for Inpatient Clinical Trials. J Diabetes Sci Technol. 2023 Nov;17(6):1527-1552. doi: 10.1177/19322968231191104. Epub 2023 Aug 17. PMID 37592726
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37592726/